CLINICAL TRIAL: NCT05266092
Title: Activation of the Contact System and the Immune System in Patients With Chronic Kidney
Brief Title: Activation of the Contact System and the Immune System in Patients With Chronic Kidney Disease.
Acronym: AKIM-CKD
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Katrine Pilely, Postdoc, Odense University Hospital
Other Study IDs: OP_1579
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Contact system; Infection; Innate immune system; Coagulation; Chronic kidney disease; Hemodialysis; End-stage renal disease
MeSH Terms: conditions — Infections; Thrombosis; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for collecting citrated and EDTA plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Participants with chronic kidney disease undergoing hemodialysis
  Interventions: Other: Observational study
- Participants with chronic kidney disease, not in dialysis
  Interventions: Other: Observational study
- Participants with chronic kidney disease undergoing peritoneal dialysis
  Interventions: Other: Observational study
- Healthy participants
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
Patients with end-stage renal disease undergoing hemodialysis (HD) are burdened with extremely high mortality rates (15% per year) and during the early stage (≤120days) the mortality rate is even higher (27% per year). Cardiovascular complications and bloodstream infections (BSIs) account for the vast majority of deaths in HD patients. In Denmark, BSIs occur in 14% of HD patients per year and is most frequently caused by Staphylococcus aureus (44%). The most frequent infectious complication is endocarditis that has fatal outcomes in ≈50% of the cases. Overall, 10% of HD patients die within 30 days after a positive blood culture for S. aureus. This project aims to answer key questions regarding HD patients' decreased ability to fight S. aureus BSIs and in particular the potential exacerbating effect of HD. We hypothesize that HD patients' blood is significantly compromised by the process of HD, to an extend that lowers immunoactivity against S. aureus. Moreover, we hypothesize, that contact activation promotes the coagulability of blood thus promoting biofilm formation by S. aureus which increases the overall risk of BSI. We will test these hypotheses by collecting blood and analyzing the inflammation and coagulation status in plasma samples from participants before and after HD. We will compare the level of the inflammatory markers in plasma from participants undergoing HD (n=180) to the level in plasma samples from three control groups: healthy volunteers (n=120), participants with renal disease not in dialysis (n=60) and participants undergoing peritoneal dialysis (n=40).

ELIGIBILITY:
Participants with chronic kidney disease undergoing hemodialysis Inclusion criteria

* Age >18 years
* Chronic kidney disease
* Hemodialysis

Exclusion criteria:

- Acute kidney disease

Participants with chronic kidney disease, not in dialysis Inclusion criteria

* Age >18 years
* Chronic kidney disease (eGFR from <15 to 44)

Exclusion criteria:

* Acute kidney disease
* Hemodialysis
* Peritoneal dialysis

Participants with chronic kidney disease undergoing peritoneal dialysis Inclusion criteria

* Age >18 years
* Chronic kidney disease
* Peritoneal dialysis

Exclusion criteria:

- Acute kidney disease

Healthy volunteers Inclusion criteria

* Age >18 years
* Blooddonors

Exclusion criteria:

- NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Blood samples and clinical information is collected from 180 participants with chronic kidney disease undergoing hemodialysis, before and after dialysis. Their levels of components from the innate immune system in plasma are compared to the levels in plasma samples from three control groups: 60 participants with chronic kidney disease not in dialysis, 60 participants with chronic kidney disease undergoing peritoneal dialysis and 120 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Plasma level of cHK | At enrollment
  cHK is the final activation product of the contact activation system

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No